CLINICAL TRIAL: NCT04564261
Title: Examining the Effectiveness of the myPlan App to Prevent Dating Violence With Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00241935; R01CE002979 (NIH)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-07

CONDITIONS: Intimate Partner Violence
Keywords: Intimate Partner Violence; Dating Violence; Relationships; Safety Planning; Adolescent; Technology; App; Teen
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myPlan Teen Group (Experimental): Personalized Healthy Relationship and Safety Planning Tool.
  Interventions: Behavioral: Personalized Healthy Relationship and Safety Planning Tool
- Usual Care Teen Control Group (Active Comparator): Usual Care Teen Relationships and Health Resource.
  Interventions: Behavioral: Usual Care Teen Relationship and Health Website

INTERVENTIONS:
Behavioral: Personalized Healthy Relationship and Safety Planning Tool — The app delivers evidence-based information and resources in three sections:
  My Relationship: contains a series of activities (e.g., "quizzes") to raise awareness of common myths about unhealthy relationships, determine characteristics of healthy relationships, examine the red flags in an unhealthy relationship, and assess risk factors for more severe abuse. Participants are provided with personalized messages about their relationship health and safety based on the answers they endorse.
  My Strategies: personalized strategies to increase participants' safety and well-being based on responses in the previous section.
  My Resources: direct links to the National Dating Abuse hotline, textline, and chatline, as well as personalized health and safety resources.
  Other Names: myPlan Teen
  Arms: myPlan Teen Group
Behavioral: Usual Care Teen Relationship and Health Website — The control group website will provide participants with tools to learn about health topics including examining healthy relationships. The resources will be targeted to adolescents. The control group website is not personalized to the participant or their relationship.
  Arms: Usual Care Teen Control Group

SUMMARY:
Intimate partner violence (IPV), including violence in teen dating relationships [teen dating violence (TDV)], is a common and a serious threat to adolescent health, safety, and well-being. TDV may include psychological/emotional abuse, sexual harassment or coercion, stalking (including cyberstalking), and physical or sexual violence. For many, the first experience of violence is in a dating or casual relationship with a partner or acquaintance during adolescence. Therefore, the objective of this study is to examine the effectiveness of an adapted version of the myPlan app for adolescents (ages 15-17 years) to prevent and respond to TDV. myPlan is an app available for mobile download or by web browser that interactively assists users to assess the health and safety of user's intimate relationship, receive personalized strategies on how build healthier relationships, stay safe and healthy while navigating an unsafe relationship, and get connected to support and resources.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 15-17 years old
* Lives in the United States
* Reports current or past 6 months physical violence, sexual violence, emotional abuse, verbal abuse, or staking (including cyberstalking or electronic aggression) by a dating/casual/intimate/ex-intimate partner
* Speaks/reads English
* Has access to a safe device (e.g., smartphone, tablet, or computer) with internet access and comfortable downloading an app or using the internet
* Has a safe contact phone number or email address

Exclusion Criteria:

* Younger than 15 years of age
* Older than 17 years of age
* Does not report current or past 6 months abuse from a dating/casual/intimate/ex- intimate partner
* Does not speak/read English
* Does not have access to a safe device (e.g., smartphone, tablet, or computer) with internet access
* Does not have a safe contact phone number or email address

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 617 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in safety behaviors measured by the Safety Behavior Checklist | Baseline, 3-, 6-, 12-months
  Percent of safety behaviors that a person has tried that they found helpful measured on checklist adapted from Intimate Partner Violence Strategies Index to assess for the range of formal and informal help seeking strategies used to halt, escape, or resist violence, and the helpfulness of each strategy.
Change from baseline in State of Change in Enacting Safety Behaviors | Baseline, 3-, 6-, 12-months
  Score on a 0 - 5 scale indicating stage a person is in with regard to taking action to make their relationship healthy with 0 indicating no action and 5 indicating full action.

SECONDARY OUTCOMES:
Change from baseline in survivors' dating abuse experience measured by Conflict in Adolescent Dating Relationships Inventory (CADRI) | Baseline, 3-, 6-, 12-months
  CADRI is an 11 item scale with a 5 point response scale (never to always) that measures the frequency of experiencing different forms of dating abuse
Change from baseline in survivors' depression measured by Pediatric Depressive Symptoms - Short Form 8a. | Baseline, 3-, 6-, 12-months
  The Pediatric Depressive Symptoms - SF 8a is an 8 items scale with a 5 point response scale (never to always) that measures the frequency of different depressive symptoms. It was developed as part of the Patient-Reported Outcomes Measurement Information System (PROMIS).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Glass, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University School of Nursing, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri